CLINICAL TRIAL: NCT02258984
Title: Can the Venus 1000 Help Clinicians Treat Patients With Severe Sepsis or Acute Heart Failure? The CVP Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mespere Lifesciences Inc. (Industry)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1407013246
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Severe Sepsis; Acute Heart Failure
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open physician access to Venus 1000 CVP data (Other)
  Interventions: Device: Mespere Venus 1000 Non-Invasive CVP System
- No open physician access to Venus 1000 CVP data (Other)
  Interventions: Device: Mespere Venus 1000 Non-Invasive CVP System

INTERVENTIONS:
Device: Mespere Venus 1000 Non-Invasive CVP System — The Venus 1000 CVP System is a non-invasive central venous pressure measurement system that utilizes the proven science of NIRS. Approved by FDA, received Health Canada Medical Device Licence and CE Marked, the Venus 1000 has been proven to be clinically equivalent to measurements made via right heart catheterization.

SUMMARY:
The purpose of this study is to evaluate the impact that the Venus 1000 non-invasive CVP system has on the management of emergency department (ED) patients with fluid sensitive conditions.

DETAILED DESCRIPTION:
The ability to non-invasively, accurately, and continuously measure CVP to assess the preload status of ED patients could lead to its inclusion into existing protocols (similar to EGDT), or the development of novel protocols for the treatment of patients with fluid sensitive conditions. The majority of other non-invasive measures of preload, such as ultrasound of the inferior vena cava or the passive leg raise technique are not continuous measures and require some type of effort or skill on the part of the clinician. Continuous methods of assessing preload include CVP measurement through a central venous catheter, esophageal Doppler monitoring, and pulse contour analysis via arterial catheter monitoring, all of which involve invasive procedures.

The Venus CVP device is non-invasive and has continuous monitoring capabilities. The data acquired from this project will allow us to determine whether emergency physicians will, in practice, utilize the information provided by a non-invasive CVP monitoring device to assist in the management of their patients with severe sepsis or acute HF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or greater
* English speaking
* Clinical diagnosis of: 1) Severe Sepsis, or 2) Acute Heart Failure

Exclusion Criteria:

* Traumatic injuries
* Active bleeding
* Pregnancy
* Prisoners
* Central venous catheter placement in the internal jugular or subclavian veins
* Bilateral external jugular vein catheterizations
* Concurrent enrollment into an interventional clinical trial that may affect subject treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
30-day Readmission | 30 days

SECONDARY OUTCOMES:
Total amount of IV fluid administered over hospitalization | 30 days
Dose, timing and duration of all IV vasoactive medications | 30 days
Length of stay in hospital | 30 days
Duration of respiratory support | 30 days
Rapid response activations | 30 days
Mortality (in hospital, 7-day, 30-day) | 30 days
Number of repeat ED visits through 30 days post-discharge | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Favot, MD, Principal Investigator — Wayne State University; Philip Levy, MD, FACEP, Principal Investigator — Wayne State University
Locations (1):
- Detroit Receiving Hospital, Detroit, Michigan, United States